CLINICAL TRIAL: NCT00539747
Title: Meaning Making Among Asymptomatic Individuals With a Positive Presymptomatic Genetic Test Result for Huntington Disease
Brief Title: Making Sense of a Positive Genetic Test Result for Huntington Disease
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908005; 08-HG-N005
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-08-05

CONDITIONS: Huntington Disease
Keywords: Presymptomatic; Huntington Disease; Meaning Making; Genetic Testing; HD
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This exploratory study will examine ways in which individuals approach a positive genetic test for Huntington Disease (HD). HD is a neurodegenerative disorder that causes emotional, cognitive, and movement problems, and currently there is no way to prevent, stop or reverse the progression of the disease. It is passed down through a mutation in a normal gene, and each child of an HD parent has a 50-50 chance of inheriting the HD gene. The study is designed to explore how individuals adjust to their new genetic status and evaluate any perceived mental or emotional barriers to that adjustment. Currently, little is known about how individuals come to terms with a positive genetic test result for a condition that has no known cure or effective treatment. The results of this study may give health care providers and counselors more information about how to help patients who are at risk for developing HD make sense of their new genetic status.

Candidates will be prescreened and referred to the study by clinics that specialize in genetic testing and counseling. Candidates must be 18 years old or older and must have received a positive genetic test result for HD at least one month prior to the study. They must also perceive themselves to be asymptomatic-that is, without existing HD symptoms.

During the study, participants will be interviewed and asked a series of questions about their decision to pursue testing, their life since the testing, and the things that they have found helpful or unhelpful since receiving the test results. The interviews will be recorded and will last approximately 60 minutes. Participants also will receive a follow-up phone call within two to three days to ensure their general psychological well-being after the interview.

DETAILED DESCRIPTION:
Huntington Disease (HD) is a progressive neurological condition, eventually leading to death. Presymptomatic, predictive genetic testing can inform individuals of their genetic status. A positive genetic test result can be a threatening event. In adapting to threatening events people often try and find meaning in the experience. Meaning making refers to the attempt to understand an event or experience and its significance in the context of one's life. The search for meaning can eventually lead to acceptance of an event or experience, and is considered an important component of adaptation. Although it has been established that testing for HD can be a significantly stressful event, and that meaning making is a frequent response towards adaptation, little is known about this process among individuals faced with a positive genetic test result for HD. This study will describe meaning making in a population of presymptomatic individuals with a positive genetic test result for HD.

Semi-structured interviews will be conducted, recorded, transcribed, and analyzed. A typology of common themes will be compiled and reported. Data gathered from these interviews will improve understanding of the phenomenon of meaning making in this population, and will contribute to the existing literature on the role of meaning making in cognitive adaptation. This study will specifically help gain insight into the process of meaning making among individuals who have tested positive for HD, and may potentially inform the ways in which health care professionals can help facilitate meaning-making among this population, in their process of adaptation to a stressful live event.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Participants for this study will be men and women, age 18 or older, who have undergone presymptomatic genetic testing for HD, received a positive test result and currently perceive themselves as being asymptomatic. To obtain a range of experiences, the investigator (PR) will attempt to recruit individuals with a range of elapsed time since their positive test result.

INCLUSION CRITERIA:

* 18 years or older
* Able to speak and understand English
* Received results that they believe are positive at least one month ago
* Perceive themselves to be asymptomatic
* Willing and able to read and describe the consent form before the phone interview

EXCLUSION CRITERIA:

* Test result less than a month ago
* Believe that they got a negative test result
* Believe themselves to be symptomatic
* Obvious symptoms of dementia or serious mental illness that would preclude consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2007-10-01; Study Completion 2008-08-05

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Daaleman TP, Frey BB, Wallace D, Studenski SA. Spirituality Index of Well-Being Scale: development and testing of a new measure. J Fam Pract. 2002 Nov;51(11):952. PMID 12485549
- [Background] Decruyenaere M, Evers-Kiebooms G, Cloostermans T, Boogaerts A, Demyttenaere K, Dom R, Fryns JP. Psychological distress in the 5-year period after predictive testing for Huntington's disease. Eur J Hum Genet. 2003 Jan;11(1):30-8. doi: 10.1038/sj.ejhg.5200913. PMID 12529703
- [Background] Bowes DE, Tamlyn D, Butler LJ. Women living with ovarian cancer: dealing with an early death. Health Care Women Int. 2002 Feb;23(2):135-48. doi: 10.1080/073993302753429013. PMID 11868961